CLINICAL TRIAL: NCT05908500
Title: Generating Evidence to Optimize Lay Rescuer Cardiopulmonary Resuscitation (CPR) Training: a Longitudinal Study of Frequency, Modality, and Design Features Impacting Skill Retention
Brief Title: Gathering Evidence on Best Practices for Lay Rescuer CPR Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Responsible Party: Principal Investigator, Lorrel Toft, Associate Professor of Medicine, University of Nevada, Reno
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Lay Rescuer CPR Training 2026
Record Dates: First submitted 2023-01-13; First posted 2023-06-18 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Arrest, Out-Of-Hospital
Keywords: Cardiopulmonary Resuscitation; cardiopulmonary resuscitation training; Lay Rescuer cardiopulmonary resuscitation; lay rescuer cardiopulmonary resuscitation training
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: Aim 1: A 4-year, cluster-randomized trial at a rural high school evaluates the impact of CPR training frequency and duration on skill retention, confidence, and emotional readiness. Students (N~1,200) are assigned by class year to different training schedules using standard, gamified, or brief refresher formats. CPR skills, knowledge, and psychosocial outcomes are assessed annually.
  Aim 2: A 2-year, individually randomized trial at a suburban high school compares four chest compression practice tools: high-fidelity manikin, low-fidelity manikin, a novel "no-head" manikin, and improvised objects. Ninth-grade students (N~432) are assessed post-training and at 1 year for CPR skill quality (rate, depth, recoil, hand placement) using objective measurement tools.
Who Masked: Outcomes Assessor
Masking Description: The statistical analysis will be masked as to which intervention subjects received, with simple "A," "B," etc. designation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Every 2 year standard CPR training (Active Comparator): Receives two 60-minute instructor-led CPR trainings: once in 9th grade and again in 11th grade
  Interventions: Behavioral: CPR Training
- Annual Standard CPR training (Active Comparator): Receives a 60-minute instructor-led CPR training each year for three years.
  Interventions: Behavioral: CPR Training
- High-Frequency, Blended Training (Active Comparator): Starts with a 30-minute serious game-based session, followed by 10-minute refreshers every semester for four years (8 total sessions).
  Interventions: Behavioral: CPR Training
- Annual Serious Game Training (Active Comparator): Receives a 30-minute serious game-based training session once per year for three years.
  Interventions: Behavioral: CPR Training
- Control (No Intervention): No CPR training
- Standard High-fidelity Manikin (Active Comparator): Uses a commercially available torso manikin with realistic chest mechanics and feedback. Serves as the gold standard comparator for CPR training.
  Interventions: Device: CPR Manikin Type
- Low-Fidelity Manikin (Active Comparator): Uses a basic inflatable torso manikin with minimal feedback or resistance. Represents a low-cost, commonly used alternative in schools and communities.
  Interventions: Device: CPR Manikin Type
- No-Head Manikin (Prototype) (Active Comparator): Uses a custom-built spring-based device with a silicone topper and realistic force-displacement properties that closely mimic the human chest. Tests whether an affordable, biomechanically accurate prototype can improve compression quality.
  Interventions: Device: CPR Manikin Type
- Non-Traditional Object (Active Comparator): Uses improvised materials (e.g., toilet paper rolls) to simulate chest compressions. Evaluates the feasibility and effectiveness of ultra-low-cost CPR practice tools
  Interventions: Device: CPR Manikin Type

INTERVENTIONS:
Behavioral: CPR Training — Various durations and frequencies of CPR training
  Arms: Annual Serious Game Training; Annual Standard CPR training; Every 2 year standard CPR training; High-Frequency, Blended Training
Device: CPR Manikin Type — Various types of CPR manikins are compared
  Arms: Low-Fidelity Manikin; No-Head Manikin (Prototype); Non-Traditional Object; Standard High-fidelity Manikin

SUMMARY:
The goal of this prospective trial is to compare CPR skill and attitudes in lay rescuers. The main question[s] it aims to answer are:

* What is the optimal training timing, duration, and frequency for lay rescuers that leads to CPR skill retention?
* What is the impact of CPR manikin type (high-fidelity, inflatable, nontraditional objects) on skill retention?
* How do specific features of training modality -- such as contextualization, gamification, and emotional engagement -- impact skill proficiency, knowledge retention, and attitudes about CPR?

Participants will

* Answer pre-training questionnaires
* Participate in CPR training
* Participate in CPR skills testing
* Answer post-training questionnaires

Researchers will compare different methods of training, different frequencies of training, and different manikin types.

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest (OHCA) remains a major public health crisis in the United States, with over 350,000 cases annually and low survival rates. Lay rescuer cardiopulmonary resuscitation (CPR) can double survival, yet widespread gaps in training access, skill retention, and emotional readiness persist. While most U.S. states mandate high school CPR training, implementation quality varies, and traditional formats have remained unchanged for over 60 years. These methods are often time-consuming, expensive, and poorly suited for adolescents, leading to low participation and rapid skill decay.

This study addresses these critical gaps by comparing various CPR training methods and procedures. The project tests the effectiveness of different training frequencies, durations, and delivery modes-including traditional instructor-led sessions, brief refreshers, and a novel, emotionally immersive serious game. The serious game leverages gamification, competition, and scenario-based learning to build "emotional muscle memory" and prepare students for real-world emergencies.

Participants are enrolled from two high schools-one rural, one suburban-and randomized by class or individual into training arms with varied schedules and compression practice tools. These tools range from high-fidelity manikins to low-fidelity devices and improvised household objects. Outcomes include CPR performance metrics (compression rate, depth, recoil, and hand placement), knowledge retention, emotional engagement (measured via validated psychometric scales), and confidence in responding to cardiac arrest.

Training sessions are delivered during the academic year, and students are assessed immediately after training and again at annual follow-up points. Data are collected in a de-identified format using school-issued ID numbers, ensuring participant confidentiality. Analysis will use generalized estimating equations and mixed-effects models to assess the impact of training method and frequency on skill retention and psychosocial readiness. The study also explores the role of contextualization, emotional engagement, and gamification as mediators of improved CPR performance.

Ultimately, this multi-year trial aims to identify scalable, cost-effective strategies that optimize CPR training outcomes for lay rescuers. By improving technical skill retention and emotional preparedness, the study addresses key priorities for public health impact and aligns with NHLBI's strategic goals to reduce mortality from sudden cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* All students at participating schools

Exclusion Criteria:

* Previous CPR training (will be included in the CPR training but excluded from analysis)
* Physical injury which prevents performing CPR
* Student or parent opt-out

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
CPR Skill Retention | 1-4 years
  High-quality CPR as measured by compression rate (per minute), depth (inches), and correct hand placement. High-quality CPR is defined as correct rate (100-120/min) AND >70% of compressions at appropriate depth (2-2.4inches) with appropriate hand placement.

SECONDARY OUTCOMES:
CPR Attitudes | 1-4 years
  Participant confidence and intention to perform CPR, measured using Likert-scale items and validated engagement questionnaires.
CPR Knowledge Retention | 1-4 years
  Percentage of correct answers on a standardized multiple-choice test assessing CPR knowledge and AED use.
Emotional Profile | 1-4 years
  Emotional responses captured by the Positive and Negative Affect Schedule (PANAS), measuring affective realism and readiness.
Learner Engagement | 1-4 years
  Subjective engagement and perceived relevance of CPR training, measured via Likert scales and the Narrative Engagement Scale.

OTHER OUTCOMES:
Training Feature Effects (Contextualization, Gamification, Emotional Impact) | 1-4 years
  Exploratory outcome assessing how specific training design elements influence CPR skills, knowledge, and self-efficacy through mediation and regression analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Lorrel Toft, Principal Investigator — University of Nevada, Reno
Locations (1):
- University of Nevada Reno, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
All data is gathered and reported in de-identified, aggregate form, per IRB and school official direction.